CLINICAL TRIAL: NCT03052426
Title: Occupational Therapy's Role in Promoting Community Wellness: A Multi-modal Approach to Combat Sedentary Behavior in the Workplace Utilizing Sit-Stand Workstations
Brief Title: Occupational Therapy's Role in Promoting Community Wellness Utilizing Sit-Stand Workstations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Brandy Brown, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1612397536
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Strain; Sedentary Lifestyle
MeSH Terms: conditions — Musculoskeletal Pain; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- 30 Minute Group (Active Comparator): This group will use the Ergotron WorkFit-TL (a sit to stand work station) and be required to alternate periods of sitting and standing every 30 minutes throughout their workday.
  Interventions: Device: Ergotron WorkFit - TL
- 60 Minute Group (Active Comparator): This group will use the Ergotron WorkFit-TL (a sit to stand work station) and be required to alternate periods of sitting and standing every 60 minutes throughout their workday.
  Interventions: Device: Ergotron WorkFit - TL
- 90 Minute Group (Active Comparator): This group will use the Ergotron WorkFit-TL (a sit to stand work station) and be required to alternate periods of sitting and standing every 90 minutes throughout their workday.
  Interventions: Device: Ergotron WorkFit - TL

INTERVENTIONS:
Device: Ergotron WorkFit - TL — A sit to stand work station.

SUMMARY:
The aim of this study is to combat the growing global health issue of sedentary behavior and the associated health consequences of prolonged sitting in the workplace. The population of desk-based workers makes up a relatively large population and are an important target for this health promoting initiative with a focus on improving posture, encouraging movement, and fostering a more active and healthy business community. It's important to recognize that occupational therapy practitioners can contribute to community health promotion/disease prevention programs by the skill-set of practitioners to understand habits and routines that influence the adoption and maintenance of healthy behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must spend > 50% of their work day seated at the computer
* Participants must be primarily English speaking
* Participants must work within the Health Sciences Center building at West Virginia University

Exclusion Criteria:

* Participants who are less than 18 years of age
* Participants who are not primarily English speaking
* Participants who spend <50% of their work day seated at the computer
* Participants who do not work within the Health Sciences Center building at West Virginia University
* Participants who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-08-27 (Actual); Study Completion 2017-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandy Brown, OTD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Groups:
- 30 Minute Group: This group will be required to alternate periods of sitting and standing every 30 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
- 60 Minute Group: This group will be required to alternate periods of sitting and standing every 60 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
- 90 Minute Group: This group will be required to alternate periods of sitting and standing every 90 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
Period: Overall Study
Arm/Group | 30 Minute Group | 60 Minute Group | 90 Minute Group
Started | 6 | 6 | 6
Completed | 4 | 5 | 5
Not Completed | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The desks were donated to the division for the purpose of research. We only received 20 desks, therefore 18 was the max number of individuals who were enrolled to allow for replacement desks to be immediately available in the event that we should need them.
Groups:
- 30 Minute Group: roup members will be required to alternate periods of sitting and standing every 30 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
- 60 Minute Group: roup members will be required to alternate periods of sitting and standing every 60 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
- 90 Minute Group: roup members will be required to alternate periods of sitting and standing every 90 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
- Total: Total of all reporting groups
Arm/Group | 30 Minute Group | 60 Minute Group | 90 Minute Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.36) | 41.67 (11.11) | 41.5 (11.15) | 45.06 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 14
  Male | 2 | 1 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 4 | 5 | 6 | 15
  Mixed | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  African American | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 0
Marital Status [Count of Participants; unit: Participants]
  Single | 1 | 3 | 1 | 5
  Cohabitating | 1 | 0 | 0 | 1
  Married | 3 | 2 | 5 | 10
  Divorced | 1 | 1 | 0 | 2
  Widowed | 0 | 0 | 0 | 0
Employment [Count of Participants; unit: Participants]
  Part-Time | 1 | 0 | 0 | 1
  Full-Time | 5 | 6 | 6 | 17
Role [Count of Participants; unit: Participants]
  Managerial | 0 | 1 | 2 | 3
  Professional | 3 | 2 | 1 | 6
  Administrative | 3 | 3 | 3 | 9
  Other | 0 | 0 | 0 | 0
Number of Days Worked Per Week [Mean (Standard Deviation); unit: number of days worked/week] — Mean number of days worked per week.
  number of days worked/week | 5 (0) | 5 (0) | 5 (0) | 5 (0)
Income [Count of Participants; unit: Participants]
  < 30K | 1 | 1 | 0 | 2
  30-60K | 0 | 0 | 1 | 1
  60-90K | 1 | 2 | 0 | 3
  90+K | 1 | 0 | 0 | 1
  Did not report | 3 | 3 | 5 | 11
Total Hours Worked Per Week [Mean (Standard Deviation); unit: hours/week] | 45.83 (10.44) | 41 (2.76) | 42.5 (4.81) | 43.11 (6.74)
Aches/Pains [Mean (Standard Deviation); unit: units on a scale] — The Cornell Musculoskeletal Discomfort Questionnaire consists of three scales that were compiled 1) aches and pains, 2) discomfort and 3) interference due to aches and pains. All three scales included 9 questions centered on the occurrence in body regions, including the neck, shoulder, upper and lower back, upper arms, forearm/wrist, hip, thigh, and knee/lower leg. Aches and Pains was on a 5 point scale, from 1) Never to 5) Several Times a Day. Higher scores indicated more problems in each of these areas.
  units on a scale | 2.54 (0.84) | 2.26 (0.55) | 2.06 (0.64) | 2.28 (0.67)
Uncomfortable from Aches/Pains [Mean (Standard Deviation); unit: units on a scale] — The Cornell Musculoskeletal Discomfort Questionnaire consists of three scales that were compiled 1) aches and pains, 2) discomfort and 3) interference due to aches and pains. All three scales included 9 questions centered on the occurrence in body regions, including the neck, shoulder, upper and lower back, upper arms, forearm/wrist, hip, thigh, and knee/lower leg. Discomfort (uncomfortable from aches and pains) was on a 4 point scale, from 0) Never to No Discomfort to 3) Very Uncomfortable. Higher scores indicated more problems in each of these areas.
  units on a scale | 1.20 (0.71) | 0.93 (0.24) | 1.07 (0.45) | 1.07 (0.49)
Aches/Pains Interfere with Work [Mean (Standard Deviation); unit: units on a scale] — The Cornell Musculoskeletal Discomfort Questionnaire consists of three scales that were compiled 1) aches and pains, 2) discomfort and 3) interference due to aches and pains. All three scales included 9 questions centered on the occurrence in body regions, including the neck, shoulder, upper and lower back, upper arms, forearm/wrist, hip, thigh, and knee/lower leg. Interference from Aches/Pains was on a 4 point scale, from 0) Not a problem to 3) Substantially interferes. Higher scores indicated more problems in each of these areas.
  units on a scale | 1.39 (0.51) | 0.90 (0.29) | 1.19 (0.46) | 1.16 (0.45)

OUTCOME MEASURES:

1. Primary Outcome: Reported Musculoskeletal Discomfort Per Group at 3 Months
Description: Three scales were compiled 1) aches and pains, 2) discomfort and 3) interference due to aches and pains. All three scales included 9 questions centered on the occurrence in body regions, including the neck, shoulder, upper and lower back, upper arms, forearm/wrist, hip, thigh, and knee/lower leg. Aches and Pains was on a 5 point scale, from 1) Never to 5) Several Times a Day. Uncomfortable was on a 4 point scale, ranging from 0) No Discomfort to 3) Very Uncomfortable. Interference was on a 4 point scale from 0) Not a problem to 3) Substantially interfered. Higher scores indicated more problems in each of these areas.
Time Frame: 3 months
Population: At this point in the study there were still 16 individuals enrolled.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 30 Minute Group | 60 Minute Group | 90 Minute Group
Number analyzed (Participants) | 6 | 6 | 4
units on a scale
  Aches and Pains | 1.43 (0.38) | 1.33 (0.12) | 1.47 (0.40)
  Uncomfortable from Aches | 0.46 (0.40) | 0.54 (0.40) | 0.89 (0.93)
  Interference | 0.50 (0.20) | 0.50 (0.20) | 0.65 (0.24)
Statistical Analysis 1: Comparison: 30 Minute Group vs 60 Minute Group vs 90 Minute Group; Wilcoxon/Kruskal-Wallis Tests and ChiSqaure analysis were completed for aches/pains at the three month time frame; Test type: Superiority; p = 0.9327, Chi-squared — p=0.05 is the threshold for statistical significance; ChiSqaure 0.1394, DF 2 for aches
Statistical Analysis 2: Comparison: 30 Minute Group vs 60 Minute Group vs 90 Minute Group; Wilcoxon/Kruskal-Wallis Tests and ChiSqaure analysis were completed for discomfort at the three month time frame; Test type: Superiority; p = 0.7523, Chi-squared — p=0.05 is the threshold for statistical significance; ChiSquare 0.5693, DF 2
Statistical Analysis 3: Comparison: 30 Minute Group vs 60 Minute Group vs 90 Minute Group; Wilcoxon/Kruskal-Wallis Tests and ChiSqaure analysis were completed for interference at the three month time frame; Test type: Superiority; p = 0.9196, Chi-squared — p=0.05 is the threshold for statistical significance; ChiSquare 0.1676, DF 2

2. Primary Outcome: Reported Musculoskeletal Discomfort Per Group at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 30 Minute Group | 60 Minute Group | 90 Minute Group
Number analyzed (Participants) | 4 | 5 | 5
units on a scale
  Aches and Pains | 1.56 (0.53) | 1.31 (0.27) | 1.53 (0.37)
  Uncomfortable from Aches | 0.64 (0.62) | 0.30 (0.23) | 0.80 (0.47)
  Interfere with Work | 0.47 (0.43) | 0.33 (0.31) | 0.62 (0.37)
Statistical Analysis 1: Comparison: 30 Minute Group vs 60 Minute Group vs 90 Minute Group; Wilcoxon/Kruskal-Wallis Tests and ChiSquare Analysis were completed; Test type: Superiority; p = 0.6316, Chi-squared — p=0.05 is the threshold for statistical significance; ChiSqaure 0.9190, DF 2
Statistical Analysis 2: Comparison: 30 Minute Group vs 60 Minute Group vs 90 Minute Group; Wilcoxon/Kruskal-Wallis Tests and ChiSqaure analysis were completed for discomfort at the six month time frame; Test type: Superiority; p = 0.2595, Chi-squared — p=0.05 is the threshold for statistical significance; ChiSqaure 2.6983, DF
Statistical Analysis 3: Comparison: 30 Minute Group vs 60 Minute Group vs 90 Minute Group; Wilcoxon/Kruskal-Wallis Tests and ChiSqaure analysis were completed for interference at the six month time frame; Test type: Superiority; p = 0.4495, Chi-squared — p=0.05 is the threshold for statistical significance; ChiSquare 1.5991, DF 2

3. Secondary Outcome: Reported Musculoskeletal Discomfort at Work at 3 Months and 6 Months All Groups Combined
Description: The Cornell Musculoskeletal Discomfort Questionnaire consists of three scales that were compiled 1) aches and pains, 2) discomfort and 3) interference due to aches and pains. All three scales included 9 questions centered on the occurrence in body regions, including the neck, shoulder, upper and lower back, upper arms, forearm/wrist, hip, thigh, and knee/lower leg. Aches and Pains was on a 5 point scale, from 1) Never to 5) Several Times a Day. Uncomfortable was on a 4 point scale, ranging from 0) No Discomfort to 3) Very Uncomfortable. Interference was on a 4 point scale from 0) Not a problem to 3) Substantially interfered. Higher scores indicated more problems in each of these areas.
Time Frame: Beginning of study, 3 months, and 6 months (end of study)
Population: Secondary to the individual group sizes being small, we decided to do an analysis of all of the groups combined to determine if the intervention made any impact on musculoskeletal discomfort with use over time.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 3 Months Results All Groups: Groups will be required to alternate periods of sitting and standing every 30, 60, or 90 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
- 6 Months Results All Groups: Group members will be required to alternate periods of sitting and standing every 30, 60, or 90 minutes utilizing their sit-stand workstation.
Arm/Group | 3 Months Results All Groups | 6 Months Results All Groups
Number analyzed (Participants) | 16 | 14
units on a scale
  Aches/Pains | 1.40 (0.30) | 1.46 (0.38)
  Uncomfortable from Aches | 0.60 (0.56) | 0.57 (0.47)
  Interfere with Work | 0.54 (0.45) | 0.48 (0.36)
Statistical Analysis 1: Comparison: 3 Months Results All Groups vs 6 Months Results All Groups; Three and six month results were combined and compared to baseline data for each of the outcome variables. Repeated measures MANOVAs with pairwise comparisons were used to examine the decrease of variables over time from time 1 to times 2 and 3; Test type: Superiority; p < 0.0001, MANOVA — Aches (F-test G-G Epsilon (1.26, 15.18) = 34.70, p < 0.0001)
Statistical Analysis 2: Comparison: 3 Months Results All Groups vs 6 Months Results All Groups; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0006, MANOVA — Uncomfortable (F-test G-G Epsilon (1.43, 17.15) = 14.39, p = 0.0006), from time 1 to times 2 and 3
Statistical Analysis 3: Comparison: 3 Months Results All Groups vs 6 Months Results All Groups; We used repeated measures MANOVAs with pairwise comparisons to examine the decrease of the variables over time. Significant differences for within subjects by time were found; Test type: Superiority; p < 0.0001, MANOVA — Interference (F-test G-G Epsilon (1.55, 18.66) = 34.09, p < 0.0001), from time 1 to times 2 and 3

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- 30 Minute Group: Group members will be required to alternate periods of sitting and standing every 30 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
- 60 Minute Group: Group members will be required to alternate periods of sitting and standing every 60 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
- 90 Minute Group: Group members will be required to alternate periods of sitting and standing every 90 minutes throughout their workday using the sit to stand workstation.
  Ergotron WorkFit - TL: A sit to stand work station.
Arm/Group | 30 Minute Group | 60 Minute Group | 90 Minute Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Number of participants per group were small creating decreased power for study results between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT03052426/Prot_SAP_000.pdf